CLINICAL TRIAL: NCT00804102
Title: Transcorneal Electrical Stimulation Therapy for Retinal Disease - A Randomized, Single-blind Pilot Study
Brief Title: Transcorneal Electrical Stimulation Therapy for Retinal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okuvision GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EST-2008
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Retinitis Pigmentosa; Macula Off; Primary Open Angle Glaucoma; Hereditary Macular Degeneration; Treated Retina Detachment; Retinal Artery Occlusion; Retinal Vein Occlusion; Non-Arthritic-Anterior-Ischemic Optic-Neuropathy; Hereditary Autosomal Dominant Optic Atrophy; Dry Age Related Macular Degeneration; Ischemic Macula Edema
Keywords: Retinitis pigmentosa; Macula off; Primary open angle Glaucoma; Hereditary Macular Degeneration; Treated Retina detachment; Retinal Artery Occlusion; Retinal Vein Occlusion,; Non-Arthritic-Anterior-Ischemic Optic-Neuropathy; Hereditary autosomal dominant Optic atrophy; dry Age-related Macular Degeneration; Ischemic Macula edema
MeSH Terms: conditions — Retinitis Pigmentosa; Glaucoma, Open-Angle; Retinal Artery Occlusion; Retinal Vein Occlusion; Optic Atrophy, Autosomal Dominant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Retinitis pigmentosa (Active Comparator)
  Interventions: Device: Transcorneal Electrical Stimulation
- Macula off (Active Comparator): condition after treatment of retinal detachment
  Interventions: Device: Transcorneal Electrical Stimulation
- Primary open angle Glaucoma (Active Comparator)
  Interventions: Device: Transcorneal Electrical Stimulation
- Hereditary Macular Degeneration (Active Comparator)
  Interventions: Device: Transcorneal Electrical Stimulation
- Treated Retina detachment (Active Comparator)
  Interventions: Device: Transcorneal Electrical Stimulation
- Retinal Artery Occlusion (Active Comparator)
  Interventions: Device: Transcorneal Electrical Stimulation
- Retinal Vein Occlusion (Active Comparator)
  Interventions: Device: Transcorneal Electrical Stimulation
- Non-Arteriitic-Anterior-Ischemic Optic-Neuropathy (Active Comparator)
  Interventions: Device: Transcorneal Electrical Stimulation
- Hereditary autosomal dominant Optic atrophy (Active Comparator)
  Interventions: Device: Transcorneal Electrical Stimulation
- dry Age-related Macular Degeneration (Active Comparator)
  Interventions: Device: Transcorneal Electrical Stimulation
- Ischemic Macula edema (Active Comparator)
  Interventions: Device: Transcorneal Electrical Stimulation
- Non-stimulated (Sham Comparator)
  Interventions: Device: DTL-electrode attached without energy

INTERVENTIONS:
Device: Transcorneal Electrical Stimulation — Neurostimulator drives Dawson-Trick-Litzkow electrode attached to patient eye. Different modi are used to stimulate patients.
  Arms: Hereditary Macular Degeneration; Hereditary autosomal dominant Optic atrophy; Ischemic Macula edema; Macula off; Non-Arteriitic-Anterior-Ischemic Optic-Neuropathy; Primary open angle Glaucoma; Retinal Artery Occlusion; Retinal Vein Occlusion; Retinitis pigmentosa; Treated Retina detachment; dry Age-related Macular Degeneration
Device: DTL-electrode attached without energy — DTL-electrode attached to patient eye receives no energy from neurostimulator. Treatment times remain the same as used for each treatment arm.
  Arms: Non-stimulated

SUMMARY:
Transcorneal stimulation may enable neurons to survive degeneration processes via enhanced secretion of neurotrophic substances and direct stimulation of neurons.

ELIGIBILITY:
Inclusion Criteria:

* Retinitis pigmentosa, Macula off, Primary open angle Glaucoma, Hereditary Macular Degeneration, Treated Retina detachment, Retinal Artery Occlusion, Retinal Vein Occlusion, Non-Arthritic-Anterior-Ischemic Optic-Neuropathy, Hereditary autosomal dominant Optic atrophy, dry Age-related Macular Degeneration, Ischemic Macula edema

Exclusion Criteria:

* Severe other disease such as non-proliferative diabetic retinopathy, exudative Age-related Macular Degeneration
* Age above 99 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
enhanced field of vision, enhanced visual acuity, lower threshold for electrical evoked phosphenes | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Florian Gekeler, MD, Prof, Principal Investigator — University-Eye-Hospital, Centre for Ophthalmology, D-72076 Tübingen, Germany

REFERENCES:
- [Result] Schatz A, Rock T, Naycheva L, Willmann G, Wilhelm B, Peters T, Bartz-Schmidt KU, Zrenner E, Messias A, Gekeler F. Transcorneal electrical stimulation for patients with retinitis pigmentosa: a prospective, randomized, sham-controlled exploratory study. Invest Ophthalmol Vis Sci. 2011 Jun 23;52(7):4485-96. doi: 10.1167/iovs.10-6932. PMID 21467183
- [Derived] Naycheva L, Schatz A, Rock T, Willmann G, Messias A, Bartz-Schmidt KU, Zrenner E, Gekeler F. Phosphene thresholds elicited by transcorneal electrical stimulation in healthy subjects and patients with retinal diseases. Invest Ophthalmol Vis Sci. 2012 Nov 1;53(12):7440-8. doi: 10.1167/iovs.12-9612. PMID 23049087